CLINICAL TRIAL: NCT06931743
Title: Research on the Application of Wrist and Ankle Electrical Stimulation Analgesia Therapy Device in Pain Management After Thyroid Surgery
Brief Title: The Application of Electrical Stimulation in Postoperative Pain Management of Thyroid Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaonan Huang (Other)
Responsible Party: Sponsor-Investigator, Xiaonan Huang, Principal Investigator, First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University
Organization: First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHEC2025-074
Record Dates: First submitted 2025-03-17; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Surgery; Electrical Stimulation; Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Device: CMNS6-1 Electronic Acupuncture Therapeutic Apparatus
- CMNS6-1 Electronic Acupuncture Therapeutic Apparatus (Experimental): CMNS6-1 Electronic Acupuncture Therapeutic Apparatus
  Interventions: Device: CMNS6-1 Electronic Acupuncture Therapeutic Apparatus

INTERVENTIONS:
Device: CMNS6-1 Electronic Acupuncture Therapeutic Apparatus — 1. The time selection of acupoint treatment is to return to the ward immediately,2 and 4 hours after surgery;
  2. Time of each stimulation: 30min;
  3. Acupoint extraction: According to the theory of wrist and ankle acupuncture and the location of pain, the upper 1 area (the ulnar margin on the little finger side and the depression of the flexor carpi ulnaris tendon) and the upper 2 area (between the palmaris longus tendon and the flexor carpi radialis on both sides) on the affected side (bilateral for total thyroidectomy) were selected as the intervention site, and the upper and lower parallel electrodes were placed in each area, and a total of 4 electrodes (8 electrodes on both sides) were placed.
  4. The parameter setting of the equipment: the frequency is set to 2Hz, the pulse width is set to 500μs, continuous wave is used, and the current intensity is the maximum tolerance of the subject's small pain threshold for 30min.
  Other Names: Experimental Arm
  Arms: CMNS6-1 Electronic Acupuncture Therapeutic Apparatus
Device: CMNS6-1 Electronic Acupuncture Therapeutic Apparatus — 1. The time selection of acupoint treatment is to return to the ward immediately,2 and 4 hours after surgery;
  2. Time of each stimulation: 30min;
  3. Acupoint extraction: According to the theory of wrist and ankle acupuncture and the location of pain, the upper 1 area (the ulnar margin on the little finger side and the depression of the flexor carpi ulnaris tendon) and the upper 2 area (between the palmaris longus tendon and the flexor carpi radialis on both sides) on the affected side (bilateral for total thyroidectomy) were selected as the intervention site, and the upper and lower parallel electrodes were placed in each area, and a total of 4 electrodes (8 electrodes on both sides) were placed.
  (4)30 minutes of ineffective microcurrent stimulation.
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy and safety of the wrist and ankle electrical stimulation analgesia therapy device in the management of analgesia after thyroidectomy by conducting clinical studies to collect data. It will also be combined with the Internet of Things technology to develop artificial intelligence equipment or applications to achieve remote monitoring and intelligent alarm, and improve the timeliness and initiative of pain management after thyroidectomy. In the future, we will further carry out a series of research work to explore the possible analgesic mechanisms through molecular biology and neurophysiology.

DETAILED DESCRIPTION:
Project Research Objectives：

1. Explore Innovative Analgesic Management Schemes after Thyroidectomy Through clinical trials and data analysis, evaluate the efficacy and safety of the wrist-ankle electrical stimulation analgesia device in post-thyroidectomy analgesia management. Explore more scientific, reasonable, and effective postoperative analgesia management schemes to provide theoretical basis and empirical support for clinical practice and promote the development and progress of pain management.
2. Achieve Remote Monitoring and Artificial Intelligence Application In the future, it will be combined with Internet of Things technology to develop artificial intelligence equipment or applications to achieve remote monitoring and intelligent alarm, improving the timeliness and proactiveness of post-thyroidectomy pain management.
3. Explore Related Analgesic Mechanisms The mechanism of the wrist-ankle electrical stimulation analgesia device in post-thyroidectomy analgesia may involve the gate control theory, the release of endogenous analgesic substances, and neural regulation, among others. In the future, we will conduct a series of research works, using molecular biology and neurophysiology methods to deeply explore the possible analgesic mechanisms.

Project Research Contents：

1. Parameter Setting and Evaluation of the Wrist-Ankle Electrical Stimulation Analgesia Device

1. Parameter setting of the wrist-ankle electrical stimulation analgesia device: Adjust the device parameters most suitable for post-thyroidectomy analgesia management and determine the corresponding acupoints, intervention timing, and intervention duration, etc.
2. Safety and effectiveness evaluation: Evaluate the safety and effectiveness of the selected device to ensure that it does not cause additional harm or risk to patients during use and can achieve the expected analgesic effect.

2. Formulation and Optimization of Analgesic Schemes

1. Individualized analgesic schemes: Develop individualized analgesic schemes based on patients' age, gender, weight, surgical scope, pain degree, and other factors.
2. Analgesic effect monitoring: Evaluate the pain degree of patients at different time points after surgery using VAS scores and other scales for quantitative assessment to monitor the analgesic effect.
3. Scheme optimization and adjustment: Adjust the analgesic scheme in a timely manner based on the monitoring results of the analgesic effect, such as adjusting the intervention time and stimulation duration, to achieve the best analgesic effect.

3. Clinical Application of the Wrist-Ankle Electrical Stimulation Analgesia Device

1. Operation training: Provide operation training for medical staff to ensure they can master the usage methods and precautions of the device proficiently.
2. Patient education: Educate patients on postoperative analgesia management, including relevant precautions, possible side effects and countermeasures, etc., to improve patients' compliance and encourage them to actively participate in their own pain management.
3. Observation of clinical application effects: Observe and record the pain degree, comfort level, adverse reactions, etc. of patients during the postoperative analgesia management process using the device, and evaluate its clinical application effect.
4. Remote monitoring and operation: Develop artificial intelligence equipment or mobile application APPs to achieve remote monitoring and operation.

4. Data Analysis and Mechanism Exploration

1. Data collection: Collect patients' pain scores, analgesic drug usage, adverse reaction rates, and preoperative and postoperative psychological evaluation scales, etc.
2. Statistical analysis: Use statistical methods to process and analyze the collected data, compare the effects of different analgesic schemes, and evaluate the effect, safety, and patient satisfaction of the wrist-ankle electrical stimulation analgesia device in post-thyroidectomy analgesia management based on the analysis results.
3. Exploration of analgesic mechanisms: Further explore the possible analgesic mechanisms through molecular biology and neurophysiology methods. For example, use neuroelectrophysiological techniques (such as EEG, EMG, etc.) to study the effects of electrical stimulation on neuronal activity, including changes in excitability, inhibition, and synchronization of neurons. Observe whether the neural activity patterns in pain-related brain regions change under the effect of electrical stimulation and how these changes affect pain perception. It is also possible to study whether electrical stimulation alleviates pain by activating the endogenous analgesic system, such as by releasing endorphins and other analgesic substances.

ELIGIBILITY:
1. Inclusion Criteria:

   * Be over 18 years of age;
   * The operation time is less than 4 hours;
   * Postoperative VAS pain score ≥3 points ;
   * Clear consciousness, able to answer questions accurately, free speech, no hearing impairment;
   * Informed consent
2. Exclusion Criteria:

   * Neck or thyroid surgery within the past ten years;
   * Menstruating, pregnant and lactating females;Those who are not satisfied with blood glucose control;
   * Skin injury or allergy; skin ulceration;
   * Past history of psychiatric disorder that met the diagnostic criteria of Diagnostic and Manual of Mental Disorders, DSM-IV;
   * Upper respiratory tract infection within 2 weeks before surgery;
   * History of implantation of pace or defibrillator;
   * Allergic to gel or intolerant to electrical stimulation;
   * History of chronic pain, pain VAS score 1 at the examination;
   * Use of sedative analgesic drugs for a long time or within 24 hours;
   * Particip in other clinical trials in the past 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain VAS score | Evaluation time: 1) the subject returned to the ward after surgery; 2) immediately after electrical stimulation; 3) Postoperative 3 hours、Postoperative 9 hours、Postoperative 15 hours、Postoperative 24 hours
  VAS (Visual Analogue Scale) scoring, namely visual analogue scoring, usually employs a straight line or ruler 10 centimeters long, with0 representing the "no pain end" and 10 representing the "most intense pain". The patient marks on the straight line according to the level of pain he or she, to indicate the intensity of pain and the degree of unpleasant psychological experience. The higher the VAS score, the more painful it is. 0 points: no pain; -3 points: mild pain; 4-6 points: moderate pain; 7-9 severe pain; 10 points: unbearable pain, namely severe pain
Pain-related measures | Preoperative and Postoperative 3 hours
  Pain-related indicators: Comparison of blood-related indicators between the control group and the intervention group of patients before and 3 hours after surgery, such as C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and interleukin (ILs).

SECONDARY OUTCOMES:
PONV classification | Postoperative 3 hours、Postoperative 9 hours、Postoperative 15 hours、Postoperative 24 hours
  The PONV score is a tool used to assess the severity of postoperative nausea and vomiting (PONV). The higher the PONV score, the severe the condition (1-4 mild, 5-6 moderate, 7-10 severe).
40-item Quality of Recovery (QoR-40) score | Postoperative 24 hours
  The QoR-40 instrument is a tool used to assess a patient's quality of recovery after surgery. In this instrument, a higher score usually means better quality of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Wrist and Ankle Electrical Stimulation Analgesia Therapy Device, Shanghai, Yangpu District, China

IPD SHARING:
Plan to Share IPD: No